CLINICAL TRIAL: NCT00914537
Title: Anal Cancer Screening Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909158; 09-C-N158
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Anal Cancer
Keywords: Anal Cancer; AIN; HPV; Cytology; HIV; HIV Positive
MeSH Terms: conditions — Anus Neoplasms; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Human immunodeficiency virus (HIV) positive adult men who have sex with men that are members of KPNC (Kaiser Permanente Northern California) and do not have a current anal cancer diagnosis.

SUMMARY:
Background:

* HIV-positive men who have sex with men (MSM) have rates of anal cancer that approach those of cervical cancer in women. However, unlike cervical cancer, there is no current recommended method of screening that could be used to detect anal precancerous lesions for the prevention of anal cancer in HIV-positive MSM.
* Infections by human papillomavirus (HPV) are the likely cause of cervical and anal precancer and cancer. Detecting the presence of HPV or related biomarkers has helped to identify women who may be at increased risk of cervical cancer; researchers believe that early detection of HPV or related biomarkers in MSM may be useful for anal cancer screening.

Objectives:

- To evaluate the effectiveness of various tests to detect cancer-causing HPV in HIV-positive men who have sex with men.

Eligibility:

- HIV-positive MSM that are interested in receiving anal screening for precancer

Design:

* HIV-positive MSM will respond to a self-administered risk factor questionnaire, and will undergo a physical exam and a high-resolution anoscopy at the participating clinic.
* The clinician will then collect to anal Pap specimens from each subject for research on HPV and related biomarkers.
* Participants will be followed annually for 2 years to collect additional health data for research follow-up.

DETAILED DESCRIPTION:
BACKGROUND:

Human immunodeficiency virus (HIV) positive men who have sex with men (MSM) are at risk of anal cancer that approaches the risk of cervical cancer for unscreened women living in developing countries. There is currently no accepted method for screening HIV positive MSM for anal precancer to reduce the morbidity and mortality due to anal cancer ; in the absence of a standard and effective screening modality, clinics often resort to anoscopy, a diagnostic procedure akin to colposcopy, and directed biopsies on all HIV positive MSM.

OBJECTIVE:

Evaluate the clinical performance of detecting carcinogenic human papillomavirus (HPV) DNA and RNA, individual carcinogenic HPV genotypes, cytogenetic markers, p16(INK4a) and Ki-67 immunocytochemistry staining, anal cytology, and combinations of these biomarkers for identifying HIV positive MSM with prevalent, 1 year cumulative, and 2 year cumulative anal precancer and cancer (histologically-confirmed greater than or equal to AIN3) using clinician-collected anal specimens at baseline.

ELIGIBILITY:

HIV positive MSM seeking anal cancer screening. Inclusion: 1) KPNC member; 2) documented HIV-positive status; 3) able and mentally competent to provide written, informed consent. Exclusion:A current diagnosis of anal cancer at enrollment.

DESIGN:

To address this need and to improve detection of anal precancer and cancer, we propose a screening cohort study of 1,000 HIV positive MSM participating in the Kaiser Permanente Northern California (KPNC) health maintenance program. Under written, informed consent, participating KPNC members will respond to a self-administered risk factor questionnaire and will undergo two anal specimen collections into liquid-based cytology (LBC) medium prior to a digital exam and high resolution anoscopy. Subjects will be asked to self-collect at home into the same LBC buffer and return their specimen in a prepared return envelope to evaluate the utility of self-collection for anal cancer screening. Subjects will be followed annually for two years to collect follow-up clinical data related to outcomes. Baseline clinician-collected specimens will be tested in a masked fashion for the following clinical biomarkers: 1) carcinogenic HPV DNA in aggregate and individual carcinogenic HPV genotypes; 2) carcinogenetic HPV RNA and HPV16/18 RNA; 3) cytogentic changes (3q, 5p, and 20q amplification); and 4) p16(INK4a) and Ki-67 immunocytochemical staining. For reference, clinician-collected specimens will be used to make LBC slides and evaluated by an expert cytopathology laboratory. We will estimate the clinical performance (sensitivity, specificity, positive and negative predictive values, and referral rates) for detection of prevalently-detected, one-year cumulative, and two-year cumulative histologically-confirmed anal precancer (anal intraepithelial neoplasia grade 3) or worse (greater than or equal to AIN3). We will test the self-collected anal specimens by the best molecular test(s) or combination of tests for detection of prevalently-detected greater than or equal to AIN3 as determined from testing the clinician-collected specimens. All MSM will undergo diagnostic procedures at all visits and independent of testing results, which will result in unbiased disease ascertainment.

ELIGIBILITY:
* 2.1 ELIGIBILITY CRITERIA:

Any male member of KPNC who is 1) identified as HIV positive through the Kaiser HIV registry, 2) 18 years or older, can provide written, informed consent, and 3) is not currently diagnosed with anal cancer (prior to enrollment).

2.2 INCLUSION CRITERIA:

HIV-positive men will be invited to participate, regardless of race and ethnicity, as described below if they meet the eligibility criteria. Other than having been diagnosed with anal cancer prior to enrollment, there will no other disease-based exclusions. Because of the high fraction of HIV-positive men are in fact MSM, we will not prescreen men for their sexual orientation.

2.3 EXCLUSION CRITERIA:

The exclusion criteria will be age less than 18, a current diagnosis of anal cancer rendered prior to enrollment, an unwillingness or inability (evident mental incapacity to understand the informed consent documents) to give informed consent.

Ages: 18 Years to 110 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human immunodeficiency virus (HIV) positive adult men who have sex with men that are members of KPNC (Kaiser Permanente Northern California) and do not have a current anal cancer diagnosis.@@@
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2009-06-02 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
High resolution anoscopy | 1 to 2 years
  Detection of AIN2 and AIN3 in high resolution anoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Kaiser Permanente, San Francisco, California, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Clark MA, Hartley A, Geh JI. Cancer of the anal canal. Lancet Oncol. 2004 Mar;5(3):149-57. doi: 10.1016/S1470-2045(04)01410-X. PMID 15003197
- [Background] Daling JR, Weiss NS, Hislop TG, Maden C, Coates RJ, Sherman KJ, Ashley RL, Beagrie M, Ryan JA, Corey L. Sexual practices, sexually transmitted diseases, and the incidence of anal cancer. N Engl J Med. 1987 Oct 15;317(16):973-7. doi: 10.1056/NEJM198710153171601. PMID 2821396